CLINICAL TRIAL: NCT05247073
Title: A Randomized Controlled Trial to Evaluate the Mostafa Maged Four-stitch Technique in Comparison With the Regular Method in Closure of the Episiotomy During Vaginal Delivery
Brief Title: Mostafa Maged Four-stitch Technique in Closure the Episiotomy During Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, rehab abdelhamid aboshama, lecturer of obstetrics and gynecology Faculty of medicine, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R 206
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Vaginal Delivery; Suture, Complication; Tear; Cervix; Hematoma; Ecchymosis
Keywords: Primigravida,; Episiotomy,; Childbirth,; Mostafa Maged; ecchymosis
MeSH Terms: conditions — Lacerations; Hematoma; Ecchymosis

STUDY DESIGN:
Intervention Model Description: 25 Patients of controlled group with routine closure of the episiotomy 25 Patients of study group with Mostafa Maged technique for closure of the episiotomy
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients of controlled group with routine closure of the episiotomy (Other): The vagina will be stitched using a continuous locking stitch and the perineal muscles and skin are repaired using approximately three or four individual stitches, each needing to be knotted separately to prevent them from dislodging.
  Interventions: Procedure: patients of controlled group with routine closure of episiotomy
- Patients of study group with Mostafa Maged technique for closure of the episiotomy (Active Comparator): The vagina will be stitched with the Mostafa Maged technique, The Mostafa Maged four-stitch technique uses absorbable vicryl threads with round needles 75 mm. The technique will prevent dead space formation, Good and tight hemostasis of the episiotomy strong approximation of the two edges of the episiotomy.
  Interventions: Procedure: The Mostafa Maged four-stitch technique fore closure of the episiotomy

INTERVENTIONS:
Procedure: patients of controlled group with routine closure of episiotomy — Perineal trauma is traditionally repaired in three stages: a continuous locking stitch is inserted to close the vaginal trauma, commencing at the apex of the wound and finishing at the level of the fourchette with a loop knot. The perineal muscles are then re-approximated with three or four interrupted sutures and finally, the perineal skin is closed by inserting continuous subcutaneous or interrupted transcutaneous stitches.
  The skin is then closed with inverted interrupted stitches placed in the subcutaneous tissue a few millimeters under the perineal skin edges (not transcutaneously).
  Arms: Patients of controlled group with routine closure of the episiotomy
Procedure: The Mostafa Maged four-stitch technique fore closure of the episiotomy — Identification of the apex of the episiotomy, then a simple suture is taken (0.5 cm) behind the apex of the episiotomy. First, the needle is inserted at the vaginal mucosa of the right edge of the episiotomy then extract the needle.
  The second stitch is inserted on the deep muscle layer of the same side (Right side) of the episiotomy cutting edge then extracting the needle.
  Then, insert the needle again on the left side of the episiotomy incision in the deep muscle layer on the left side of the episiotomy incision directing the tip of the needle upwards parallel to the second stitch taken.
  The fourth step is inserting the needle in the vaginal mucosa of the left side parallel to the first stitch. Continue suturing the episiotomy incision continuously in the same way till reaching the remnant of the hymen.
  Then suture the superficial perineal muscle in a continuous manner and the skin in a subcuticular manner as well.
  Arms: Patients of study group with Mostafa Maged technique for closure of the episiotomy

SUMMARY:
Most primigravida is confronted with episiotomy during childbirth to prevent the perineal and vaginal lacerations which could be performed at birth. There are many types of episiotomy which are median, mediolateral, and J-shaped episiotomy.

Prevention of the formation of the dead space during the repair of episiotomy so avoiding hematoma formation in the episiotomy area after child-birth.

The Mostafa Maged four-stitch technique uses absorbable vicryl threads with round needles 75 mm.

DETAILED DESCRIPTION:
Methodology: This technique will be applied to all women with episiotomy at the time of delivery or having tears in the perineum or the vagina. The technique uses absorbable vicryl threads with round needles 75 mm long. The technique includes the vaginal epithelium and the deep muscle layer together continuously at the same sutures. Assessment of the perineal area in the next twenty-four hours till discharge looking for (edema - hematoma - septic wound - continence - ecchymosis - dyspareunia).

ELIGIBILITY:
Inclusion Criteria:

1. Primigravida patients having episiotomies or tears in the vagina
2. Age between 18 to 40 years old

Exclusion Criteria:

1. Smokers
2. Diabetics
3. Morbidly obese patients
4. Chronic diseases such as renal diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Heamostasis of the episiotomy | 4 weeks after delivery
  Bleeding from the epistiomy or heamatoma at the epistomy
No edema at the site of episiotomy | 4 weeks after delivery
  Swelling or ecchymosis and edema at the edges of episiotomy
No infection at the episiotomy | 4 weeks after delivery
  Redness,hotness and bad odour of vaginal discharge

SECONDARY OUTCOMES:
Sexual dysfunction (pain during sexual intercourse) | 4 weeks after delivery
  Pain during sexual intercourse
Anorectal dysfunction | 4 weeks after delivery
  Inability to control passage of stool or flatus or both

CONTACTS AND LOCATIONS:
Overall Officials: Laila E Abdelfattah, Ass. prof, Principal Investigator — Associated professor of obestatrics and gynecology Faculty of medicine Fayoume university

IPD SHARING:
Plan to Share IPD: No